CLINICAL TRIAL: NCT02789293
Title: Glaucoma Treatment Using Focused Ultrasound in Open Angle Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EyeTechCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETC-EU-BN02
Record Dates: First submitted 2016-05-24; First posted 2016-06-02 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2019-07

CONDITIONS: Glaucoma
Keywords: Glaucoma; Ultrasound; Ciliary body
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Focused Ultrasound treatment (Experimental): Ultrasound ciliary pasty (UCP) using focused ultrasound
  Interventions: Device: EyeOP1 device

INTERVENTIONS:
Device: EyeOP1 device — Ultrasound Ciliary Plasty (UCP procedure) using Focused Ultrasound

SUMMARY:
The purpose of the this study is to collect safety and efficacy data on Focused Ultrasound treatment (UCP procedure) in open angle glaucoma patients without previous glaucoma surgery.

ELIGIBILITY:
Inclusion Criteria:

* Open Angle Glaucoma patient (Primary Open Angle Glaucoma (POAG) including Pigmentary Glaucoma (PG) and PseudoExfoliative Glaucoma (PXF))
* Any patients without previous conventional glaucoma surgery failure (trabeculectomy, Deep Sclerectomy, Ahmed valve, drainage device implantation, cyclo cryotherapy, Diode laser cyclo-destruction)
* Subjects where the IOP is not adequately controlled with glaucoma medication, with IOP ≥ 21 mm Hg and <30 mmHg
* No previous intraocular surgery or laser treatment during the 90 days before HIFU Day
* Age > 18 years and < 90 years
* Patient able and willing to complete postoperative follow-up requirements

Exclusion Criteria:

* Patient who has been diagnosed for normal tension glaucoma
* Ocular or retrobulbar tumor
* Ocular infection within 14 days prior to the HIFU procedure
* Ocular disease other than glaucoma that may affect assessment of visual acuity and/or IOP (choroidal hemorrhage or detachment, lens subluxation, thyroid ophthalmopathy, proliferative diabetic retinopathy, clinically significant macular edema…)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Efficacy endpoint : Reduction of intraocular pressure | 24 months
  Reduction of intraocular pressure at 24 months relative to the preoperative value assessed at each follow-up visits with the final measurement of success at 24 months

SECONDARY OUTCOMES:
Safety : rate of per and post-operative complications/adverse effects | 24 months
  rate of per-operative device and /or procedure related adverse events and post-operative complications at each follow-up visits
Efficacy endpoint : Mean IOP (mmHg) | 24 months
  Evolution of the Mean IOP (mmHg) at each visit during the follow-up period (Baseline to 24 months)
Efficacy Endpoint : Mean IOP variation (%) | 24 months
  Mean IOP variation (%) at each visit during the follow-up period
Mean Number of ocular hypotensive medications | 24 months
  Mean number of ocular hypotensive medication at each visit during the followup period

CONTACTS AND LOCATIONS:
Locations (4):
- UZ Leuven - University Hospital, Leuven, Belgium
- The Sam Rothberg Glaucoma Center, Goldschleger EyeInstitute, Sheba Medical Center, Tel Litwinsky, Israel
- Cisanello Hospital, Pisa, Italy
- Santa Maria Hospital - Faculty of Medicine of Lisbon, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No